CLINICAL TRIAL: NCT03109366
Title: Flexible Collaborative Networks and Patient-provider Partnerships in Health Care: Critical Factors
Brief Title: Electronic Tool for Interaction Between Patients and Health Professionals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: University of Oslo (Other); University Hospital of North Norway (Other); Balsfjord Municipality (Unknown); Marshfield Clinic Research Foundation (Other); Columbia University (Other); Norwegian Centre for Integrated Care and Telemedicine (Unknown)
Responsible Party: Principal Investigator, Cornelia Ruland, Professor, Oslo University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 201512/S10
Record Dates: First submitted 2011-06-24; First posted 2017-04-12 (Actual); Last update posted 2017-04-12 (Actual); Status verified 2017-04

CONDITIONS: Chronic Illness
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Online self-management support (Other): Access to online self-management support tool for six months
  Interventions: Behavioral: Online patient-provider communication service

INTERVENTIONS:
Behavioral: Online patient-provider communication service

SUMMARY:
This project's overall objective is to contribute to knowledge and innovation needed to advance ICT-arenas for timely, secure and seamless collaboration between chronically ill patients and appropriate levels of care. The investigators will expand an Internet solution that has successfully supported online patient-provider communication into a device- independent mobile, multifunctional ICT platform, called Connect 2.0, to support individually tailored collaborative care between patients and care providers on the continuum of primary-specialist care. The results will contribute to Norway's Collaboration Reform. Integrating theories from health and ICT related sciences, the project is organized into five work packages that focus on two of VERDIKTs research themes: social networking and mobile internet. We will summarize (1) the current state of collaborative health care models and their utilization of ICT research and innovations; explore challenges related to (2) information exchange between devices, platforms and systems; (3) human-computer interaction, (4) data security and confidentiality; and (5) factors related to successful adoption and implementation of Connect 2.0 patient-provider collaborative care. Finally the investigators will explore how Connect 2.0 impacts interactions, communication and organizational processes in collaborative "real world" care.

Specifically this study will:

1. Summarize the current state of collaborative health care models and their utilization of ICT research and innovations.
2. Explore challenges and propose solutions for adapting a mobile multifunctional ICT platform (Connect 2.0) into the technical and organizational infrastructures of collaborative health care.
3. Through user-centred design methods address challenges related to human computer interaction and usability of Connect 2.0.
4. Explore challenges and feasible solutions that safeguard data security and confidentiality when connecting an Internet solution with a protected health net while ensuring safe and efficient data transfer through heterogeneous networks.
5. Explore factors related to successful adoption and implementation of Connect 2.0 in real world collaborative care. Based on the above: explore impacts of a test version of Connect 2.0 on interactions, communication and organizational processes.

The work expands partnerships between the Centre for research-based innovation (SFI) consortium (7 business / research partners) called Tromsø Telemedicine Laboratory (TTL), the Norwegian Telemedicine Center (NST), the Center for Shared Decision Making and Nursing Research (CSDM) at Oslo University Hospital, the Department of Computer Science, University of Oslo, the University Hospital of Northern Norway (UNN), Balsfjord Municipality, the Biomedical Information Research Center at the Marshfield Clinic Research Foundation, and the Department of Biomedical informatics at Columbia University in New York.

ELIGIBILITY:
Inclusion Criteria:

* Chronic illness
* Receive municipal health services
* Internet access at home

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-05; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Patterns of intervention use | 6 months
  Frequency of intervention use

CONTACTS AND LOCATIONS:
Overall Officials: Cornelia M Ruland, PhD, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Rikshospitalet,, Oslo, Norway

REFERENCES:
- [Result] Mirkovic J, Kaufman DR, Ruland CM. Supporting cancer patients in illness management: usability evaluation of a mobile app. JMIR Mhealth Uhealth. 2014 Aug 13;2(3):e33. doi: 10.2196/mhealth.3359. PMID 25119490